CLINICAL TRIAL: NCT01081262
Title: A GCIG Intergroup Multicenter Phase III Trial of Open Label Carboplatin and Paclitaxel +/- NCI-Supplied Agent: Bevacizumab (NSC #704865) Compared With Oxaliplatin and Capecitabine +/- Bevacizumab as First Line Chemotherapy in Patients With Mucinous Epithelial Ovarian or Fallopian Tube Cancer (MEOC)
Brief Title: Carboplatin and Paclitaxel or Oxaliplatin and Capecitabine With or Without Bevacizumab as First-Line Therapy in Treating Patients With Newly Diagnosed Stage II-IV or Recurrent Stage I Epithelial Ovarian or Fallopian Tube Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02516; NCI-2011-02516 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0241; CDR0000667089; GOG-0241 (Other: NRG Oncology); GOG-0241 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Borderline Ovarian Mucinous Tumor; Ovarian Mucinous Cystadenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Stage IA Fallopian Tube Cancer AJCC v6 and v7; Stage IA Ovarian Cancer AJCC v6 and v7; Stage IB Fallopian Tube Cancer AJCC v6 and v7; Stage IB Ovarian Cancer AJCC v6 and v7; Stage IC Fallopian Tube Cancer AJCC v6 and v7; Stage IC Ovarian Cancer AJCC v6 and v7; Stage IIA Fallopian Tube Cancer AJCC v6 and v7; Stage IIA Ovarian Cancer AJCC V6 and v7; Stage IIB Fallopian Tube Cancer AJCC v6 and v7; Stage IIB Ovarian Cancer AJCC v6 and v7; Stage IIC Fallopian Tube Cancer AJCC v6 and v7; Stage IIC Ovarian Cancer AJCC v6 and v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Capecitabine; Carboplatin; Oxaliplatin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (carboplatin and paclitaxel) (Experimental): Patients receive carboplatin IV over 30-60 minutes on day 1 and paclitaxel IV over 3 hours on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm II (oxaliplatin and capecitabine) (Experimental): Patients receive oxaliplatin IV over 2-6 hours on day 1 and capecitabine PO BID on days 1-14. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Other: Laboratory Biomarker Analysis; Drug: Oxaliplatin; Other: Quality-of-Life Assessment
- Arm III (carboplatin, paclitaxel, bevacizumab) (Experimental): Patients receive carboplatin and paclitaxel IV as in arm I and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab IV over 30-90 minutes alone on day 1. Treatment repeats every 3 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm IV (oxaliplatin, capecitabine, bevacizumab) (Experimental): Patients receive oxaliplatin and capecitabine as in arm II, and bevacizumab as in arm III.
  Interventions: Biological: Bevacizumab; Drug: Capecitabine; Other: Laboratory Biomarker Analysis; Drug: Oxaliplatin; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm III (carboplatin, paclitaxel, bevacizumab); Arm IV (oxaliplatin, capecitabine, bevacizumab)
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
  Arms: Arm II (oxaliplatin and capecitabine); Arm IV (oxaliplatin, capecitabine, bevacizumab)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm I (carboplatin and paclitaxel); Arm III (carboplatin, paclitaxel, bevacizumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
  Arms: Arm II (oxaliplatin and capecitabine); Arm IV (oxaliplatin, capecitabine, bevacizumab)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm I (carboplatin and paclitaxel); Arm III (carboplatin, paclitaxel, bevacizumab)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies carboplatin given together with paclitaxel with or without bevacizumab to see how well it works compared with oxaliplatin given together with capecitabine with or without bevacizumab as first-line therapy in treating patients with newly diagnosed stage II-IV, or recurrent (has come back) stage I epithelial ovarian or fallopian tube cancer. Drugs used in chemotherapy, such as carboplatin, paclitaxel, oxaliplatin, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, may block tumor growth in different ways by targeting certain cells. It is not yet known which regimen of combination chemotherapy given together with or without bevacizumab is more effective in treating epithelial ovarian cancer or fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if capecitabine and oxaliplatin reduces the death rate compared to carboplatin and paclitaxel in women with mucinous adenocarcinoma of the ovary or fallopian tube.

II. To determine if bevacizumab reduces the death rate compared to no bevacizumab in women with mucinous adenocarcinoma of the ovary or fallopian tube.

SECONDARY OBJECTIVES:

I. To determine if capecitabine and oxaliplatin increases the duration of progression-free survival (PFS) compared to carboplatin and paclitaxel in women with mucinous adenocarcinoma of the ovary or fallopian tube.

II. To determine if bevacizumab increases the duration of PFS compared to no bevacizumab in women with mucinous adenocarcinoma of the ovary or fallopian tube.

III. To compare the response rates for capecitabine and oxaliplatin versus carboplatin and paclitaxel in patients with mucinous adenocarcinoma of the ovary or fallopian tube with measurable disease after initial tumor reductive surgery.

IV. To compare the response rates for bevacizumab versus no bevacizumab in patients with mucinous adenocarcinoma of the ovary or fallopian tube with measurable disease after initial tumor reductive surgery.

V. To determine the nature and degree of toxicity of capecitabine and oxaliplatin compared with that of carboplatin and paclitaxel in this cohort of patients.

VI. To determine the nature and degree of toxicity of bevacizumab in this cohort of patients.

VII. To compare capecitabine and oxaliplatin versus carboplatin and paclitaxel with respect to changes in patient reported neurotoxicity.

VIII. To determine the impact on quality of life (QOL, as measured by the Functional Assessment of Cancer Therapy-Ovarian [FACT-O] Trial Outcome Index [TOI]) following treatment with the above regimens.

TERTIARY OBJECTIVES:

I. To collect fixed and/or frozen tissue and whole blood for future research studies.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive carboplatin intravenously (IV) over 30-60 minutes on day 1 and paclitaxel IV over 3 hours on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive oxaliplatin IV over 2-6 hours on day 1 and capecitabine orally (PO) twice daily (BID) on days 1-14. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive carboplatin and paclitaxel IV as in arm I and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab IV over 30-90 minutes alone on day 1. Treatment repeats every 3 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.

ARM IV: Patients receive oxaliplatin and capecitabine as in arm II, and bevacizumab as in arm III.

After completion of study treatment, patients are followed up at 4-6 weeks, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of mucinous adenocarcinoma of the ovary or fallopian tube with either optimal (=< 1 cm residual disease) or suboptimal residual disease following initial surgery; patients may have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or no measurable disease
* All patients must have had appropriate surgery including appendectomy (unless patient has history of prior appendectomy) for ovarian or fallopian tube carcinoma with appropriate tissue available for histologic evaluation to confirm diagnosis and stage
* Patients must have stage II-IV disease (new or recurrent-chemonaïve; no brain metastasis) or recurrent stage I disease (chemonaïve)
* Newly diagnosed patients must begin protocol therapy within 10 weeks of primary debulking; for stage I recurrent patients (chemonaïve), they should begin protocol therapy within 14 days of randomization
* Patients must have a negative colonoscopy within 1 year of enrolling in the study
* Absolute neutrophil count (ANC) >= 1,500/mcl
* White blood cell (WBC) count >= 3,000/mcl
* Platelets >= 100,000/mcl
* Hemoglobin (Hgb) >= 10 g/dl (can be post transfusion)
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN) OR creatinine clearance > 50 cc/min
* Bilirubin =< 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) =< to 2.5 x ULN
* Alkaline phosphatase =< to 2.5 x ULN
* Neuropathy (sensory and motor) =< Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* Urine dipstick for proteinuria < 2+; if urine dipstick is >= 2+, 24 hour urine must demonstrate =< 1 g protein in 24 hours OR patients must have a urine protein-to-creatinine ratio (UPCR) < 1.0 mg/dL
* Prothrombin time (PT) =< 1.5 x ULN
* Activated prothrombin time (APTT) =< 1.5 x ULN
* Patients of childbearing potential must agree to practice an effective form of birth control during study treatment and for six months after completion of treatment
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients with Gynecologic Oncology Group (GOG) performance grade of 0, 1 or 2
* Patients with life expectancy > 3 months

Exclusion Criteria:

* Patients with known colon cancer or history of colon cancer
* Patients with primary peritoneal carcinoma
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last 5 years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received chemotherapy, radiotherapy or any investigational treatment for a gynecologic cancer (does include breast cancer) or colorectal cancer prior to enrollment
* Patients with a major surgical procedure anticipated during the course of the study; this includes but is not limited to: abdominal surgery (laparotomy or laparoscopy) such as colostomy or enterostomy reversal, interval or secondary cytoreductive surgery, or second look surgery; please consult with the study chair prior to patient entry for any questions related to the classification of surgical procedures
* Patients may have minor surgical procedures (i.e., mediport insertion) fine needle aspiration or core biopsies as long as it is performed > 7 days prior to the first date of bevacizumab therapy and there is no evidence of wound disruption or impaired healing
* Patients with surgery (including open biopsy) within 4 weeks prior to anticipated first dose of bevacizumab (allowing for fact that bevacizumab can be omitted from first cycle of chemotherapy)
* Patients with a history of abdominal fistula or perforation within the past 12 months
* Patients with a current, serious, non-healing wound, ulcer, or bone fracture; patients with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require weekly wound examinations
* Patients with known hypersensitivity to Chinese hamster cell products or other recombinant human or humanized antibodies
* Patients with mixed epithelial ovarian cancer histology
* Patients with tumors of low malignant potential
* History or evidence of upon physical examination of central nervous system (CNS) disease, including history of primary brain tumor or any history of brain metastases, or seizures not controlled with standard medical therapy
* Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 100 mm Hg; patients with a history of hypertension are permitted
* Myocardial infarction or unstable angina within 12 months of the first date of bevacizumab therapy
* New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication; women who have received prior treatment with anthracycline (including doxorubicin and/or liposomal doxorubicin) and have an ejection fraction < 50% will be excluded from the study
* Grade 1, category 2 or greater, peripheral vascular disease; patient cannot have anything worse than mild, symptomatic claudication with exercise
* History of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of bevacizumab therapy
* History of pulmonary embolism or deep vein thrombosis in the past 6 months
* Previous history of malabsorption or other conditions preventing oral treatment
* Patients who are pregnant or nursing
* Patients with acute hepatitis or active infection that requires parenteral antibiotics
* Patients with active bleeding or pathologic conditions that carry a high risk of bleeding such as a known bleeding disorder, coagulopathy or tumor involving the major vessels
* Patients taking warfarin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10-12 (Actual); Primary Completion 2015-02-25 (Actual); Study Completion 2026-03-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David M Gershenson, Principal Investigator — NRG Oncology
Locations (248):
- United States (248):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Wilma Chan Highland Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Pikeville Medical Center, Pikeville, Kentucky
  - Cancer Center of Acadiana, Lafayette, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 12 October 2010 and closed to patient accrual on 28 October 2013.
Period: Overall Study
Arm/Group | Arm I (Carboplatin and Paclitaxel) | Arm II (Oxaliplatin and Capecitabine) | Arm III (Carboplatin, Paclitaxel, Bevacizumab) | Arm IV (Oxaliplatin, Capecitabine, Bevacizumab)
Started | 13 | 13 | 13 | 11
Completed | 13 | 13 | 13 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and Treated Patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Carboplatin and Paclitaxel) | Arm II (Oxaliplatin and Capecitabine) | Arm III (Carboplatin, Paclitaxel, Bevacizumab) | Arm IV (Oxaliplatin, Capecitabine, Bevacizumab) | Total
Number analyzed (Participants) | 13 | 13 | 13 | 11 | 50
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 2 | 1 | 0 | 1 | 4
  30-39 years | 1 | 3 | 3 | 2 | 9
  40-49 years | 2 | 1 | 1 | 3 | 7
  50-59 years | 3 | 7 | 5 | 3 | 18
  60-69 years | 2 | 1 | 3 | 1 | 7
  70-79 years | 2 | 0 | 1 | 1 | 4
  80-89 years | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 13 | 11 | 50
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death, or the date of last contact.
Time Frame: Up to five years
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Carboplatin and Paclitaxel) | Arm II (Oxaliplatin and Capecitabine) | Arm III (Carboplatin, Paclitaxel, Bevacizumab) | Arm IV (Oxaliplatin, Capecitabine, Bevacizumab)
Number analyzed (Participants) | 13 | 13 | 13 | 11
months | 37.6 [8.8 to NA] — Upper limit not yet reached | 27.8 [9.3 to NA] — Upper limit not yet reached | 27.7 [4.9 to 53.6] | 55.7 [9.9 to NA] — Upper limit not yet reached.

2. Secondary Outcome: Participants With Grade 1 or Higher Non-serious Adverse Effects Assessed by CTCAE Version 4.0
Description: Grade 1 or higher non-serious adverse events were graded by CTC AE v 4.
Time Frame: Every cycle while on treatment, up to 5 years
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Carboplatin and Paclitaxel) | Arm II (Oxaliplatin and Capecitabine) | Arm III (Carboplatin, Paclitaxel, Bevacizumab) | Arm IV (Oxaliplatin, Capecitabine, Bevacizumab)
Number analyzed (Participants) | 13 | 13 | 13 | 11
Participants
  Abnormal lab values | 8 | 10 | 10 | 10
  Allergic reaction | 3 | 1 | 0 | 4
  Allergic rhinitis | 0 | 1 | 1 | 1
  Alopecia | 11 | 1 | 9 | 5
  Anemia | 12 | 7 | 4 | 6
  Bleeding | 1 | 1 | 3 | 5
  Cold-like symptoms | 2 | 3 | 7 | 6
  Constipation | 3 | 4 | 7 | 9
  Diarrhea | 5 | 6 | 5 | 8
  dyspnea | 2 | 1 | 3 | 0
  Edema Limbs | 0 | 1 | 0 | 0
  Fatigue | 10 | 10 | 8 | 11
  Fever | 3 | 0 | 2 | 1
  Hand/Foot Syndrome | 1 | 0 | 0 | 7
  Headache | 3 | 4 | 5 | 4
  Hypertension | 3 | 8 | 9 | 10
  Hypomagnesemia | 1 | 0 | 2 | 0
  Infection | 4 | 0 | 3 | 3
  Laryngeal Spasm | 0 | 4 | 0 | 0
  Low Lymphocytes | 1 | 1 | 2 | 0
  Low Mood | 1 | 2 | 1 | 1
  Low Neutrophils | 7 | 5 | 4 | 7
  Low platelets | 8 | 3 | 5 | 7
  Low white Blood Cells | 5 | 5 | 4 | 6
  Mucositis | 1 | 1 | 1 | 3
  Nausea/Vomiting | 8 | 8 | 9 | 9
  Oral Problems | 3 | 2 | 4 | 9
  Other | 4 | 4 | 7 | 7
  Other GI Problems | 8 | 6 | 7 | 6
  Pain | 9 | 6 | 7 | 7
  Peripheral/Sensory Neuropathy | 11 | 11 | 8 | 10
  Pneumothorax | 0 | 1 | 0 | 0
  Raised CA19-9 | 0 | 0 | 2 | 0
  Raised Blood Counts | 1 | 1 | 0 | 1
  Rash | 4 | 2 | 3 | 4
  Stomatitis | 0 | 2 | 1 | 0
  Taste Alteration | 3 | 2 | 1 | 2
  Urinary Problems | 1 | 0 | 1 | 2
  Vaginal Bleeding | 0 | 1 | 1 | 2
  Weight Gain | 0 | 1 | 1 | 2
  Weight Loss | 2 | 3 | 4 | 5

3. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria in Solid Tumors criteria (RECIST v1.0) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Is measured from date of randomization until first indication of progression based on RECIST criteria or death from any cause, or if progression-free at last contact, the date of last disease assessment up to 10 years.
Population: All Randomized Patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Carboplatin and Paclitaxel) | Arm II (Oxaliplatin and Capecitabine) | Arm III (Carboplatin, Paclitaxel, Bevacizumab) | Arm IV (Oxaliplatin, Capecitabine, Bevacizumab)
Number analyzed (Participants) | 13 | 13 | 13 | 11
Months | 36.1 [2.0 to NA] — Upper limit not yet reached | 7.4 [4.5 to NA] — Upper limit not yet reached | 15.4 [4.9 to NA] — Upper limit not yet reached | 23.3 [9.1 to NA] — Upper limit not yet reached

4. Secondary Outcome: Objective Tumor Response
Description: Complete and Partial Tumor Response by RECIST 1.1. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v.1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR),.>=30% decrease in the sum of the longest diameter of target lesions; Overall response (OR) = CR + PR
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle for the first 6 months; then every 3 months x 2; then every 6 months thereafter until disease progression, and any other time clinically indicated, up to 5 years
Population: All randomized patients with measurable disease
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm I (Carboplatin and Paclitaxel) | Arm II (Oxaliplatin and Capecitabine) | Arm III (Carboplatin, Paclitaxel, Bevacizumab) | Arm IV (Oxaliplatin, Capecitabine, Bevacizumab)
Number analyzed (Participants) | 9 | 11 | 7 | 5
Percentage of Participants | 22 [3 to 60] | 27 [6 to 61] | 43 [10 to 82] | 40 [5 to 85]

5. Secondary Outcome: Patient Reported Neurotoxicity
Description: Patient reported neurotoxicity symptoms as measured with the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - neurotoxicity subscale (short version) (FACT/GOG-Ntx subscale). The FACT/GOG-Ntx subscale contains 4 items. Each item was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). For the negative items, reversal was performed prior to score calculation. According to the FACIT measurement system, the Ntx score was the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the scale. The Ntx score ranges 0-16 with a large score suggests less neurotoxicity.
Time Frame: baseline (pre-treatment), pre cycle 4, post cycle 6, six months post-chemo, end of bevacizumab [BEV] (or 39 weeks after completion of chemotherapy in the non-BEV arms or in those who discontinue BEV), six months after BEV, and years 2, 3, 4, and 5
Population: Patients who provided a valid FACT/GOG-Ntx subscale assessment. Data were not collected at certain time points for certain arms.
Measure: Mean (Standard Deviation); unit: units on a scale.
Arm/Group | Arm I (Carboplatin and Paclitaxel) | Arm II (Oxaliplatin and Capecitabine) | Arm III (Carboplatin, Paclitaxel, Bevacizumab) | Arm IV (Oxaliplatin, Capecitabine, Bevacizumab)
Number analyzed (Participants) | 3 | 3 | 3 | 5
units on a scale.
  Baseline (pre-treatment) | 16.0 (0.0) | 15.3 (1.2) | 14.3 (2.9) | 16.0 (0.0)
  Pre-cycle 4 | 7.3 (4.2) | 11.8 (5.3) | 12.7 (3.5) | 5.7 (4.9)
  Post cycle 6 | 6.5 (2.1) | 11.7 (4.0) | 11.0 (5.6) | 8.0 (6.3)
  Six months post chemo: number analyzed (Participants) | 3 | 0 | 3 | 5
  Six months post chemo | 5.0 (4.2) |  | 11.3 (5.7) | 10.7 (2.3)
  End of bevacizumab (BEV): number analyzed (Participants) | 1 | 1 | 3 | 5
  End of bevacizumab (BEV) | 16.0 (NA) — Standard deviation is not presented if only one valid assessment was received. | 10.0 (NA) — Standard deviation is not presented if only one valid assessment was received. | 9.5 (4.9) | 11.7 (3.8)
  Six months after BEV: number analyzed (Participants) | 1 | 1 | 3 | 5
  Six months after BEV | 10.0 (NA) — Standard deviation is not presented if only one valid assessment was received. | 10.0 (NA) — Standard deviation is not presented if only one valid assessment was received. | 9.0 (4.2) | 7.0 (9.9)
  2 years after BEV: number analyzed (Participants) | 1 | 1 | 3 | 1
  2 years after BEV | 8.0 (NA) — Standard deviation is not presented if only one valid assessment was received. | 14.0 (NA) — Standard deviation is not presented if only one valid assessment was received. | 5.5 (4.9) | 16.0 (NA) — Standard deviation is not presented if only one valid assessment was received.
  3 years after BEV: number analyzed (Participants) | 1 | 0 | 3 | 1
  3 years after BEV | 14.0 (NA) — Standard deviation is not presented if only one valid assessment was received. |  | 9.5 (4.9) | 16.0 (NA) — Standard deviation is not presented if only one valid assessment was received.
  4 years after BEV: number analyzed (Participants) | 0 | 0 | 3 | 0
  4 years after BEV |  |  | 6.5 (6.4) |
  5 years after BEV: number analyzed (Participants) | 0 | 0 | 3 | 0
  5 years after BEV |  |  | 7.5 (3.5) |

6. Secondary Outcome: Patient Reported Quality of Life
Description: Patient reported quality of life was measured with the Treatment Outcome Index of the Functional Assessment of Cancer Therapy for endometrial cancer (FACT-O TOI). The FACT-O TOI is a scale for assessing general QOL of ovarian cancer patients. It consists of three subscales: Physical Well Being (7 items), Functional Well Being (7 items), and Ovarian Cancer subscale (11 items). Each item in the FACT-O TOI was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). For the negative statements (or questions), reversal was performed prior to score calculation. According to the FACIT measurement system, a subscale score was the summation of the individual item scores if more than 50% of subscale items were answered. The FACT-O TOI score ranges 0-100 with a large score suggests better QOL
Time Frame: as for outcome 5
Population: All Randomized Patients with at least one post-baseline QOL assessment reported were averaged. Data were not collected at certain time points for certain arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Carboplatin and Paclitaxel) | Arm II (Oxaliplatin and Capecitabine) | Arm III (Carboplatin, Paclitaxel, Bevacizumab) | Arm IV (Oxaliplatin, Capecitabine, Bevacizumab)
Number analyzed (Participants) | 3 | 3 | 3 | 5
units on a scale
  Baseline (pre-treatment) | 62.6 (12.6) | 62.3 (29.5) | 68.7 (9.7) | 75.4 (15.9)
  Pre-Cycle 4 | 57.5 (4.8) | 72.9 (16.4) | 68.7 (2.1) | 76.0 (12.5)
  Post-Cycle 6 | 65.2 (4.0) | 73.5 (9.1) | 68.3 (5.5) | 71.8 (14.1)
  Six Months Post-Chemo: number analyzed (Participants) | 3 | 0 | 3 | 5
  Six Months Post-Chemo | 74.1 (14.2) |  | 80.3 (12.2) | 68.7 (29.7)
  End of Bevacizumab (BEV): number analyzed (Participants) | 1 | 1 | 3 | 5
  End of Bevacizumab (BEV) | 68.9 (NA) — Standard deviation is not presented if only one valid assessment was received. | 53.3 (NA) — Standard deviation is not presented if only one valid assessment was received. | 73.0 (22.6) | 49.9 (31.4)
  Six Months after BEV: number analyzed (Participants) | 1 | 1 | 3 | 5
  Six Months after BEV | 54.0 (NA) — Standard deviation is not presented if only one valid assessment was received. | 53.0 (NA) — Standard deviation is not presented if only one valid assessment was received. | 87.5 (7.8) | 70.5 (26.2)
  2 Years after BEV: number analyzed (Participants) | 1 | 1 | 3 | 1
  2 Years after BEV | 71.7 (NA) — Standard deviation is not presented if only one valid assessment was received. | 56.0 (NA) — Standard deviation is not presented if only one valid assessment was received. | 76.3 (15.2) | 77.0 (NA) — Standard deviation is not presented if only one valid assessment was received.
  3 Years after BEV: number analyzed (Participants) | 1 | 0 | 3 | 1
  3 Years after BEV | 76.4 (NA) — Standard deviation is not presented if only one valid assessment was received. |  | 80.5 (17.7) | 76.0 (NA) — Standard deviation is not presented if only one valid assessment was received.
  4 Years after BEV: number analyzed (Participants) | 0 | 0 | 3 | 0
  4 Years after BEV |  |  | 71.5 (24.7) |
  5 Years after BEV: number analyzed (Participants) | 0 | 0 | 3 | 0
  5 Years after BEV |  |  | 78.0 (17.0) |

7. Other Pre Specified Outcome: Numbers and Percentages of Patients With Mutations in the Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) Oncogene
Description: Will be tabulated. Interactions between the mutational status of the KRAS oncogene and treatment will be examined.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Study treatment and up to 5 years after treatment discontinuation
Arm/Group | Arm I (Carboplatin and Paclitaxel) | Arm II (Oxaliplatin and Capecitabine) | Arm III (Carboplatin, Paclitaxel, Bevacizumab) | Arm IV (Oxaliplatin, Capecitabine, Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 3/13 | 4/13 | 2/13 | 3/11
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13 | 13/13 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Carboplatin and Paclitaxel) (N=13) | Arm II (Oxaliplatin and Capecitabine) (N=13) | Arm III (Carboplatin, Paclitaxel, Bevacizumab) (N=13) | Arm IV (Oxaliplatin, Capecitabine, Bevacizumab) (N=11)
Allergic reaction (Immune system disorders) | 1 | 1 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Bleeding (General disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Fever (General disorders) | 1 | 0 | 0 | 0
GI perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Low Neutrophils (Investigations) | 1 | 0 | 1 | 0
Low Platelets (Investigations) | 1 | 0 | 0 | 0
Nausea/Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 1
Peripheral/sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Thromboembolic Event (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Carboplatin and Paclitaxel) (N=13) | Arm II (Oxaliplatin and Capecitabine) (N=13) | Arm III (Carboplatin, Paclitaxel, Bevacizumab) (N=13) | Arm IV (Oxaliplatin, Capecitabine, Bevacizumab) (N=11)
Laryngeal Spasm (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0
Low Lymphocytes (Investigations) | 0 | 1 | 1 | 0
Low Mood (Psychiatric disorders) | 1 | 2 | 1 | 1
Low Neutrophils (Investigations) | 7 | 5 | 4 | 7
Low platelets (Investigations) | 8 | 3 | 5 | 7
Low White Blood Cells (Investigations) | 5 | 5 | 4 | 6
Mucositis (General disorders) | 1 | 1 | 1 | 3
Nausea (Gastrointestinal disorders) | 8 | 8 | 9 | 9
Oral problems (Gastrointestinal disorders) | 3 | 2 | 4 | 9
Other (General disorders) | 4 | 4 | 7 | 7
Other GI Problems (Gastrointestinal disorders) | 8 | 6 | 7 | 7
Pain (General disorders) | 9 | 6 | 7 | 7
Peripheral/sensory Neuropathy (Nervous system disorders) | 11 | 11 | 8 | 10
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Raised CA19-9 (Investigations) | 0 | 0 | 2 | 0
Raised Blood counts (Investigations) | 1 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 3 | 4
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Taste Alteration (Nervous system disorders) | 3 | 2 | 1 | 2
Urinary Problems (Renal and urinary disorders) | 1 | 0 | 1 | 2
Vaginal Bleeding (Reproductive system and breast disorders) | 0 | 1 | 1 | 2
Weight Gain (Investigations) | 0 | 1 | 1 | 2
Weight Loss (Investigations) | 2 | 3 | 4 | 5

LIMITATIONS AND CAVEATS:
The majority of patients were deemed not to have primary mucinous ovarian cancer post hoc. The trial accrued slowly and was stopped early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less